CLINICAL TRIAL: NCT01548378
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety and Efficacy of NL003 in Subject With Critical Limb Ischemia
Brief Title: Safety and Efficacy Study Using Gene Therapy for Critical Limb Ischemia
Acronym: NL003CLI-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Northland Biotech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL003CLI-II
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Arterial Occlusive Disease; Ulcers; Ischemia; Peripheral Vascular Disease
Keywords: HGF; Gene; Critical Limb Ischemia
MeSH Terms: conditions — Arterial Occlusive Diseases; Ulcer; Ischemia; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Dose (Experimental): Patients in this treatment group will receive 8mg NL003 respective in D0、14、28
  Interventions: Genetic: NL003
- Middle Dose (Experimental): Patients in this treatment group will receive 6mg NL003 respective in D0、14、28
  Interventions: Genetic: NL003
- Low Dose (Experimental): Patients in this treatment group will receive 4mg NL003 in D0、14、28
  Interventions: Genetic: NL003
- Placebo (Placebo Comparator): Patients in this group will receive normal saline respective in D0、14、18
  Interventions: Other: Normal Saline

INTERVENTIONS:
Genetic: NL003 — Day 0: 8mg of NL003 (32 injections of 0.5ml of NL003) Day 14: 8mg of NL003 (32 injections of 0.5ml of NL003) Day 28: 8mg of NL003 (32 injections of 0.5ml of NL003)
  Other Names: HGF plasmid; pCK-HGF-X7
  Arms: High Dose
Genetic: NL003 — Day 0: 6mg of NL003 (24 injections of 0.5ml of NL003) and 4ml normal saline(8 injections) Day 14: 6mg of NL003 (24 injections of 0.5ml of NL003) and 4ml normal saline(8 injections) Day 28: 6mg of NL003 (24 injections of 0.5ml of NL003) and 4ml normal saline(8 injections)
  Other Names: HGF plasmid; pCK-HGF-X7
  Arms: Middle Dose
Genetic: NL003 — Day 0: 4mg of NL003 (16 injections of 0.5ml of NL003) and 8ml normal saline(16 injections) Day 14: 4mg of NL003 (16 injections of 0.5ml of NL003) and 8ml normal saline(16 injections) Day 28: 4mg of NL003 (16 injections of 0.5ml of NL003) and 8ml normal saline(16 injections)
  Other Names: HGF plasmid; pCK-HGF-X7
  Arms: Low Dose
Other: Normal Saline — Day 0: 16ml of Normal Saline (32 injections ) Day 14: 16ml of Normal Saline (32 injections ) Day 28: 16ml of Normal Saline (32 injections )
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether intramuscular injections of NL003 into the calf is safe and effective in the treatment of critical limb ischemia

DETAILED DESCRIPTION:
Management of CLI process consumes a significant amount of healthcare resources,and the new therapeutic approaches are required.

Hepatocyte growth factor (HGF) has been shown to be a potent angiogenic growth factor stimulating the growth of endothelial cells and migration of vascular smooth muscle cells. Because of its pluripotent capabilities, increasing the availability of HGF in ischemic tissues to achieve therapeutic angiogenesis has been a growing area of research.

This study will use NL003, which is a DNA plasmid that contains novel genomic cDNA hybrid human HGF coding sequence (HGF-X7) expressing two isoforms of HGF, HGF 728 and HGF 723. As there are currently no approved drugs that can reverse CLI and as most patients have exhausted surgical and endovascular intervention options, inducing angiogenesis in the affected limb with NL003 may result in an increase in tissue perfusion, which, in turn improve wound healing, reduce pain and improve limb salvage rates.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 30 and 80years of age
* Diagnosis of critical limb ischemia(ASO、TAO、DAO)，Rutherford Class 4 or 5, including:

  * A resting ankle systolic pressure of ≤ 70 mmHg in the affected limb; or
  * A resting toe systolic pressure of ≤ 50 mmHg in the affected limb; or
  * For patients in which measurement of ankle systolic pressure is not feasible , TcPO2 ≤ 30mmHg; Only unilateral affected limb receive treatment。
* Significant stenosis (≥ 75%) of one or more of the following arteries:

superficial femoral, popliteal as verified by angiography（DSA、CTA、MRA） within 12 months prior to enrollment

* Be willing to maintain current drug therapy for peripheral arterial disease throughout the course of the study
* Be willing to maintain ulcer treatment
* Be willing to infertility throughout the course of the study
* If the subject is of child-bearing potential, she must have a negative urine pregnancy test result prior to study enrollment
* Tumor screening result is no clinic meaning，including:
* Signing the informed consent document prior to being subjected to any study related procedures

Exclusion Criteria:

* Subjects who have undergone a successful revascularization procedure or sympathectomy within 12 weeks prior to study entry.
* Acute advanced CLI
* Subjects that will require an amputation in the target leg within 4 weeks, or significant stenosis (≥ 75%) of Aortoiliac
* Subjects with evidence of active infection or deep ulceration exposing bone or tendon in the extremity planned for treatment
* Heart Failure with a NYHA classification of III or IV
* Stroke、myocardial infarction or unstable angina within last 3 months
* Uncontrolled hypertension defined as sustained systolic blood pressure (SBP) > 180 mmHg or diastolic BP (DBP) > 110 mmHg
* Ophthalmologic conditions pertinent to proliferative retinopathy or conditions that preclude standard ophthalmologic examination
* Can not correctly describe the symptoms and feeling
* Subjects with advanced liver disease including decompensated cirrhosis, jaundice, ascites or bleeding varices
* Subjects currently receiving immunosuppressive medications chemotherapy, or radiation therapy
* Positive HIV,active Hepatitis B(determined by HBsAb\ HBcAb\HBsAg) or C infection
* Specific laboratory values at Screening including: Hemoglobin < 8.0 g/dL, WBC < 3,000 cells per microliter, platelet count <75,000/mm3, AST and/or ALT > 3 times the upper limit of normal or any other clinically significant lab abnormality which in the opinion of the investigator should be exclusionary
* Elevated PSA unless prostate cancer has been excluded
* Patients with a recent history (< 5 years) of or new screening finding of malignant neoplasm except basal cell carcinoma or squamous cell carcinoma of the skin (if excised and no evidence of recurrence); patients with family history of colon cancer in any first degree relative are excluded unless they have undergone a colonoscopy in the last 12 months with negative findings
* Subjects requiring > 100 mg daily of acetylsalicylic acid,COX-2 inhibitor drug(s) or high dose steroids (excepting inhaled steroids)
* Subjects with any co- morbid conditions likely to interfere with assessment of safety or efficacy or with an estimated life expectancy of less than 12 months
* History of drug or alcohol abuse / dependence in the past 12 months
* Use of an investigational drug or treatment in past 3 months

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The difference in ulcer area between baseline and the D180. | Day180
  Rutherford 5 only
The difference in pain level between baseline and the D180 as determined by VAS | Day 180

SECONDARY OUTCOMES:
Change in tissue oxygenation (TcPO2) from baseline to D180 | Day0、14、28、60、90、180
Difference in percentage of pain level decreased by 50% determined by VAS from baseline to D180 | Day0、14、28、60、90、180
Difference in percentage of ulcer area decreased by 50% from baseline to D180 | Day0、14、28、60、90、180
Difference in ABI and TBI from baseline to D180 | Day0、14、28、60、90、180
Difference in QOL score (VascuQol) from baseline to D180 | Day0、14、28、60、90、180
Percentage of ulcer complete healing | Day180
Situation of ulcer healing | Day180
Ulcer healing after gangrene treatment | Day180
Major amputation rate | Day180

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Shijitan Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality
  - Wuhan Union Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning

REFERENCES:
- See also: Related Info — http://www.northland-bio.com/